CLINICAL TRIAL: NCT01940692
Title: TOPICAL AND INTRAVENOUS ADMINISTRATION OF TRANEXAMIC ACID ARE EQUALLY EFFECTIVE IN DIRECT ANTERIOR TOTAL HIP ARTHROPLASTY - A PROSPECTIVE RANDOMIZED CONTROLLED TRIAL
Brief Title: Topical and Intravenous Administration of TXA Are Equally Effective in DAA THA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Jacobs Brecht, Medical student, Ziekenhuis Oost-Limburg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TXA01
Record Dates: First submitted 2013-08-28; First posted 2013-09-12 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Osteoarthrosis
MeSH Terms: conditions — Osteoarthritis | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous tranexamic acid (Active Comparator): Will receive 1.5g intravenous tranexamic acid preoperatively
  Interventions: Drug: 1.5g intravenous Exacyl
- Intra-articular tranexamic acid (Experimental): Will receive 3g intra-articular tranexamic acid after wound closing
  Interventions: Drug: 3.0g intra-articular Exacyl

INTERVENTIONS:
Drug: 1.5g intravenous Exacyl — intravenous administration of 1.5g Exacyl preoperatively
  Arms: Intravenous tranexamic acid
Drug: 3.0g intra-articular Exacyl — 3g Intra-articular Exacyl administration postoperatively
  Arms: Intra-articular tranexamic acid

SUMMARY:
Through a randomized controlled trial, we will compare the intravenous administration of tranexamic acid with the intra-articular application after a total hip arthroplasty through direct anterior approach.

* RCT, prospective study
* Academic-monocentric study
* Clinical outcome measurements The postoperative blood loss will be the primary outcome. Secondary outcomes are

  1. The rate of perioperative and postoperative blood transfusion
  2. The number of blood units transfused
  3. The length of hospital stay
  4. Perioperative given intravenous isotonic fluid

The Null-hypothesis is that there is no significant difference in postoperative blood loss between intra-articular and intravenous administration of TXA.

DETAILED DESCRIPTION:
Study protocol:

Topical application of tranexamic acid compared to the intravenous administration in total hip arthroplasty with the direct anterior approach A prospective, randomized, clinical trial

Researchers: B. Jacobs and Dr. S. Ghijselings Supervisors: Dr. R. Driesen, Dr. M. Beran, Dr. R. Heylen Coördinerend supervisor: Prof dr. K. Corten

Background

The prevalence of total hip arthroplasty (THA) is increasing and the accompanied blood loss cannot be overlooked. In 2007, 17,347 patients underwent THA in Belgium and that number grows every year by an average of 2.9%. The average amount of blood loss associated with THA was ranging from 1000 to 2000mL. Therefore the substantial perioperative blood loss frequently necessitates blood transfusion. Although complications have decreased, morbidity and high costs due to blood transfusion still exist.

To avoid blood transfusion after THA, tranexamic acid (TXA) can be administered. TXA, a synthetic amino acid that blocks the lysine binding sites on plasminogen in a competitive way, is an antifibrinolytic agent. TXA can be administered intravenously or intra-articular. The ideal method of providing TXA remains topic of debate. Several studies have proven that intravenous application reduces blood loss and the need for blood transfusion in patients undergoing THA . In contrast, after intravenous administration only a small percentage of the drug reaches the target location, the rest distributes across the whole body. Hence the risk of possible side effects after intravenous administration, like thromboembolic events and gastrointestinal complaints, theoretically is greater.

Local application of TXA could get around these possible systemic side effects. The benefit of topical application of TXA has been proven for dental surgery, cardiac surgery, spine surgery and total knee arthroplasty. In a case-control study, Van Elst et al (20) recently proved that local application of TXA after THA reduces total bleeding by 100 to 380 mL in comparison to placebo.

Null - Hypothesis

In this study, we will compare the efficacy of intra-articular application of TXA to the intravenous administration in terms of postoperative blood loss.

Our hypothesis is that there is no significant difference in postoperative blood loss between intra-articular and intravenous administration of TXA.

Materials and Methods

What:

* Power analysis
* RCT, prospective study
* Monocentric study
* Clinical outcome measurements Each patient will give written consent for inclusion in the study. This prospective, single-centered, randomized clinical trial is designed to enroll a total of 120 patients who meet the inclusion criteria, with approximate 60 patients in each group. Patients are allocated to a) intravenous application of TXA or b) intra-articular administration of TXA, with use of a computer-generated randomization table.

Inclusion criteria:

All adults (patients over the age of eighteen years) who were scheduled for a primary unilateral total hip arthroplasty due to osteoarthritis at Ziekenhuis Oost-Limburg, Genk, Belgium are eligible for inclusion in the study.

Exclusion criteria:

A patient is excluded from the study if he or she has a history of coagulopathy, allergy to tranexamic acid, preoperative anemia, fibrinolytic disorders, history of arterial or venous thromboembolic disease, disturbances of color vision, pregnancy, breastfeeding, major comorbidities and participation in another clinical trial.

Preoperative protocol

With a blood sample, preoperative hemoglobin level will be measured. This hemoglobin level is used to calculate postoperative blood loss.

Surgical procedure

Spinal anesthesia will be given to all patients and standard monitoring will be used during surgery.

Two orthopedic surgeons (K.C. and R.D.) participated in this study. Both surgeons use the same surgical technique, the direct anterior approach (DAA). The type of prosthesis used will be based on the surgeon's preference and patient age, activity level and demands. All implants are cementless and a surgical drain is placed to collect the postoperative blood loss.

Whenever intraoperative surgical, medical, or anesthetic complications occur, TXA will not be administered and the patient will be excluded from the study. Prophylaxis antibiotic, 2g of cephalosporin, will be intravenously administered right before the intervention and this is repeated three times within 24 hours over a constant time interval.

Tranexamic acid procedure

To ensure the double-blinding upset of this study, the 60 patients from the control group receive a solution of 1.5g TXA in 100ml 0.9%NaCl, administered intravenously before closure of the incision. A dose of 3g TXA is applied intra-articular to the other group of 60 patients. The intra-articular injection is applied after THA, when the wound already has been closed. Two hours after wound closing, the surgical drain will be opened. The two hour wait after wound closing is proven most successful.

Postoperative follow-up

Postoperative applied prophylaxis and early mobilization will be used to prevent deep-vein thrombosis (DVT). The administered prophylaxis include daily low molecular weight heparin until six weeks after surgery. While in the hospital, patients will be examined daily for any clinical symptoms of DVT. Patients also receive compressive stockings to wear after surgery.

Postoperative hemoglobin levels are measured at the first and the fourth day postoperative. All patients remained in the hospital for a minimum of 5 days.

Outcome measures

The primary outcome is the postoperative blood loss. The difference between total blood loss and intraoperative blood loss is used to predict the postoperative blood loss for each patient.

The secondary outcomes includes:

1. The rate of perioperative and postoperative blood transfusion
2. The number of blood units transfused
3. The length of hospital stay
4. Perioperative given intravenous isotonic fluid

The criterion for the transfusion of blood products is a hemoglobin level of <8.0 g/dL if the patient developed intolerable symptoms of anemia or any comorbidities that may have been related to anemia and was not attributable to another cause or ongoing blood loss was occurring. If transfusion is necessary, the amount of units of packed red blood cells is estimated according to the hemoglobin level or the severity of symptoms with the intention to increase the hemoglobin level to 8.0 g/dL.

Statistical analysis

Each patient will receive a detailed brochure with information concerning the study procedure and a written informed consent will be obtained.

Patients can decline the offer for participation in the study. In that case these patients shall get treatment as proposed. Patients that accept to participate are randomized to either the group of intravenous administration or intra-articular administration of tranexamic acid. These patients will receive a number and will be randomly assigned to either the intravenous or intra-articular group by computer.

ELIGIBILITY:
Inclusion Criteria:

* All adults (patients over the age of eighteen years) who were scheduled for a primary unilateral total hip arthroplasty due to osteoarthritis at Ziekenhuis Oost-Limburg, Genk, Belgium are eligible for inclusion in the study.

Exclusion Criteria:

* History of coagulopathy
* Allergy to tranexamic acid
* preoperative anemia
* fibrinolytic disorders
* history of arterial or venous thromboembolic disease
* disturbances of color vision
* pregnancy
* breastfeeding
* major comorbidities
* participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Postoperative Bloodloss | Day 1 after surgery
  Measured with a simple blood sample on day one after surgery

SECONDARY OUTCOMES:
Rate of perioperative and postoperative blood transfusion | Patients will be followed for the duration of hospital stay, an expected average of 5 days
Number of blood units transfused | Patients will be followed for the duration of hospital stay, an expected average of 5 days
Length of hospital stay | Measured when patient goes home, minimum 5 days after surgery
Severity of pain at rest as determined with use of a visual analog scale | Patients will be followed for the duration of hospital stay, an expected average of 5 days
  possible range 0 to 10
Perioperatively given intravenous isotonic fluid | Patients will be followed for the duration of hospital stay, an expected average of 5 days
  Done for calculation of the factor dilution after surgery

OTHER OUTCOMES:
Preoperative hemoglobin level | The day before the surgery
  Measured with a simple blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Kristoff Corten, Prof. dr., Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

REFERENCES:
- [Derived] Vles GF, Corten K, Driesen R, van Elst C, Ghijselings SG. Hidden blood loss in direct anterior total hip arthroplasty: a prospective, double blind, randomized controlled trial on topical versus intravenous tranexamic acid. Musculoskelet Surg. 2021 Dec;105(3):267-273. doi: 10.1007/s12306-020-00652-0. Epub 2020 Mar 10. PMID 32152813
- See also: Main site of department of orthopedics in Ziekenhuis Oost-Limburg — http://www.orthopediegenk.be/nl
- See also: Site of hospital Ziekenhuis Oost-Limburg — http://www.zol.be